CLINICAL TRIAL: NCT00111397
Title: A Study of Adjuvant Cytokine Therapy in Pulmonary Mycobacterium Avium Complex and Other Pulmonary Nontuberculous Mycobacterial Infections
Brief Title: Adjuvant Cytokine Therapy to Treat Pulmonary Mycobacterium Avium Complex Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050156; 05-I-0156
Record Dates: First submitted 2005-05-19; First posted 2005-05-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-08-04

CONDITIONS: Mycobacterium Avium-Intracellulare Infection
Keywords: Mycobacterial; Interferon; GM-CSF; Microarray; Proteomics; Mycobacterium Avium Complex Infection; MAC
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection | interventions — Interferon-gamma; Granulocyte-Macrophage Colony-Stimulating Factor

INTERVENTIONS:
Procedure: Cytokine therapy
Drug: Interferon Gamma, GM-CSF

SUMMARY:
Mycobacterium avium complex (MAC) are ubiquitous organisms that cause isolated pulmonary disease in otherwise healthy patients with yet undefined susceptibilities. Patients typically present with a history of chronic cough, eventually progressing to hemoptysis, fever, and hypoxia. With half or more of all patients failing standard three-drug therapy, this is an insidious disease with a poor prognosis. Under the natural history protocol of nontuberculous mycobacterial infection (NTM; #01-I-0202), 46 patients with diagnosed pulmonary MAC disease are being studied. Numerous studies have suggested that a dysregulation in cytokine production may make these patients susceptible to mycobacterial infection. Cytokines are particularly important in the activaction of macrophages, which help to clear mycobacterial infection. Interferon gamma 1b (Actimmune) and GM-CSF (Leukine) are two cytokine therapies that have been approved in the treatment of chronic granulomatous disease and post-transplantation hematopoietic reconstitution, respectively. A number of in vitro studies suggest that either or both of these therapies may help to clear MAC infection. Given the poor outcomes of therapy and the persistent, debilitating nature of the disease, new therapies are desperately needed, and many are being tried without benefit of scientific foundation. Currently, there are no prospective trials that show any effect of these drugs in the lung delivered subcutaneously. This protocol proposes to perform a pilot study to evaluate the effects, if any, of these macrophage stimulating cytokines in the context of ongoing pulmonary MAC infection.

Aims:

To determine the local and systemic effect, if any, of adjuvant IFN gamma and GM-CSF in pulmonary MAC patients.

Methods:

Fifteen patients will be randomized into three treatment groups of five patients each. The first group will receive a standard drug regimen, based on the 1997 ATS guidelines. The second and third groups, in addition to receiving the standard therapy, will also receive three months of (IFN{gamma}) and GM-CSF, respectively. All patients will undergo bronchoscopy with bronchoalveolar lavage (BAL) at the beginning of the study, after three months, and at six months.

In addition to obtaining traditional subjective and objective clinical measures, both proteomic and genomic analysis of the BAL will be performed to determine if cytokine therapy effects any detectable change in the lungs. In vitro studies on typ...

DETAILED DESCRIPTION:
Mycobacterium avium complex (MAC) and other pulmonary nontuberculous mycobacteria (P-NTM) are ubiquitous organisms that cause isolated pulmonary disease in otherwise healthy patients with yet undefined susceptibilities. Patients typically present with a history of chronic cough, eventually progressing to hemoptysis, fever, and hypoxia. With half or more of all patients failing standard three-drug therapy, this is an insidious disease with a poor prognosis. Under the natural history protocol of nontuberculous mycobacterial infection (NTM; #01-I-0202), 46 patients with diagnosed pulmonary MAC disease, 20 patients with M. abscessus disease, and 14 with other types of mycobacteria (M. fortuitum, M. massiliense, M. mucogenicum and M. chelonae) are being studied.

Numerous studies have suggested that a dysregulation in cytokine production may make these patients susceptible to mycobacterial infection. Cytokines are particularly important in the activation of macrophages, which help to clear mycobacterial infection. Interferon gamma 1b (Actimmune) and GM-CSF (Leukine) are two cytokine therapies that have been approved in the treatment of chronic granulomatous disease and post-transplantation hematopoietic reconstitution, respectively. A number of in vitro studies suggest that either or both of these therapies may help to clear MAC infection. Given the poor outcomes of therapy and the persistent, debilitating nature of the disease, new therapies are desperately needed, and many are being tried without benefit of scientific foundation. Currently, there are no prospective trials that show any effect of these drugs in the lung delivered subcutaneously. This protocol proposes to perform a pilot study to evaluate the effects, if any, of these macrophage stimulating cytokines in the context of ongoing pulmonary mycobacterial infection.

Aims:

To determine the local and systemic effect, if any, of adjuvant IFN gamma and GM-CSF in P-NTM patients.

Methods:

Fifteen patients will be randomized into three treatment groups of five patients each. The first group will receive a standard drug regimen, based on the 1997 ATS guidelines. The second and third groups, in addition to receiving the standard therapy, will also receive three months of (IFN{gamma}) and GM-CSF, respectively. All patients will undergo bronchoscopy with bronchoalveolar lavage (BAL) at the beginning of the study, after, after three months, and at six months.

In addition to obtaining traditional subjective and objective clinical measures, both proteomic and genomic analysis of the BAL will be performed to determine if cytokine therapy effects any detectable change in the lungs, In vitro studies on type II alveolar macrophages culled from these patients before and after cytokine therapy will also be performed.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for this protocol, a patient must meet the following five criteria:

Diagnosed with M. avium complex (MAC) lung disease or other pulmonary mycobacterial infection based on the 1997 version of American Thoracic Society (ATS) diagnostic criteria and have positive AFB smear or culture for mycobacterial infection at least three months prior to the date of enrollment. Patients with only histological evidence of mycobacterial infection without positive smear or culture will not qualify for this protocol even if they meet the ATS diagnostic criteria for nontuberculous mycobacterial lung infection.

A patient must have radiographic evidence on high resolution computerized tomography of changes that are consistent with pulmonary mycobacterial infection. These include, but are not limited to: multiple small nodules (less than 5 mm), and cylindrical bronchiectasis.

The patient must be on a treatment regimen based on ATS guidelines that has been stable for at least three months. By stable, we mean that the patient has been tolerating the regimen without any significant adverse reactions, and that no new agents have been begun in the last three months.

The patient must be female and can be post-menopausal (either through natural menopause or surgical removal of her ovaries) or menstruating. If the patient is still menstruating and randomized to a study group receiving a cytokine she must agree to monthly pregnancy testing, while on study, as well as to utilizing a barrier type of contraception or abstinence. She must not be under 40 years of age at the time of enrollment in the study.

The patient must be enrolled in protocol # 01-I-0202 ("Natural History, Genetics, Phenotype, and Treatment of Non-Tuberculoid Mycobacterial Infections").

EXCLUSION CRITERIA:

Patients with pulmonary MAC disease who do not meet the above entry criteria.

Patients with any of the following preexisting medical conditions:

1. HIV positive
2. asthma
3. active cancer requiring treatment
4. hepatic disease (defined as either a history of cirrhosis, or grade 3 or 4 hepatic toxicity by the Toxicity Table in Appendix II of protocol)

Patients who are unable to tolerate bronchoscopy. This will be defined by the following criteria:

1. A pulse oximetry reading less than 100% when given supplemental oxygen at 100% FiO2.
2. Clinically significant reactive airway disease that does not respond to bronchodilators.

Patients with the following laboratory abnormalities:

1. creatinine greater than 1.5 mg/dL
2. Hemoglobin less than 9 mg/dL
3. WBC less than 3,000
4. Platelets less than 150,000
5. ALT greater than 82 U/L, or AST greater than 78 U/L.
6. Bilirubin greater than 2.0 mg/dL
7. Alkaline phosphates greater than 232 U/L

Patients with a preexisting allergy or history of allergic reactions to study or protocol medications. These include, but are not necessarily limited to: IFN-gamma, GM-CSF, azithromycin/ clarithromycin, ethambutol, rifampin/ rifabutin, anesthetic agents employed in bronchoscopy, or any yeast-derived products.

Patients who are unable to maintain the described follow up schedule. Likewise, patients who are unable to give informed consent are excluded from the study.

Patients with clinical diagnosis of cystic fibrosis.

Patients who are either currently smoking, or have a previous history of smoking that exceeds 20 pack years.

Patients with prior treatment with either IFN-gamma or GM-CSF within the last three months.

Patients with known history of cardiac, endocrine, neurologic or other medical conditions that the principal investigator deems dangerous or unsuitable for enrollment will be excluded.

Patients who are either pregnant or lactating. Also, menstruating patients who are randomized to a study group receiving a cytokine and refuse to use appropriate barrier forms of contraception or abstinence during this trial be excluded.

Patients who, at any time during this trial, have an active lung infection caused by either Staphylococcus or a gram negative rod are excluded from this trial until this infection has been successfully treated.

Patients that need to use supplemental oxygen.

Patients who have a Forced Vital Capacity less than 40% predicted.

Patients who are unable to walk and participate in the 6MWT.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2005-05-13; Primary Completion 2010-08-04 (Actual); Study Completion 2010-08-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Prince DS, Peterson DD, Steiner RM, Gottlieb JE, Scott R, Israel HL, Figueroa WG, Fish JE. Infection with Mycobacterium avium complex in patients without predisposing conditions. N Engl J Med. 1989 Sep 28;321(13):863-8. doi: 10.1056/NEJM198909283211304. PMID 2770822
- [Background] Iseman MD, Buschman DL, Ackerson LM. Pectus excavatum and scoliosis. Thoracic anomalies associated with pulmonary disease caused by Mycobacterium avium complex. Am Rev Respir Dis. 1991 Oct;144(4):914-6. doi: 10.1164/ajrccm/144.4.914. PMID 1928970
- [Background] Chalermskulrat W, Gilbey JG, Donohue JF. Nontuberculous mycobacteria in women, young and old. Clin Chest Med. 2002 Sep;23(3):675-86. doi: 10.1016/s0272-5231(02)00010-2. PMID 12371003